CLINICAL TRIAL: NCT00296296
Title: Randomized Open Label Study Comparing the Metabolic Control of Kidney Transplant Recipients With Type 2 Diabetes Receiving Either Prograf or Neoral as Part of a ATG Induction, Prednisone Free and Monitored MMF Immunosuppressive Regimen.
Brief Title: Immunosuppression Impact on the Metabolic Control of Kidney Transplant With Pre-Existing Type 2 Diabetes (DM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephan Busque, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95442
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Kidney Transplant; Diabetes Mellitus, Type 2; Diabetic Nephropathy
Keywords: kidney Transplant; Type II Diabetes; Diabetic Nephropathy; Immunosuppression; Cyclosporin; Tacrolimus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Cyclosporine; Tacrolimus; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporin (Active Comparator): Patients receive cyclosporin (dose-adjusted to pre-established targets) as immunosuppressive calcineurin inhibitor (CNI) and Diabetes Education / Management (therapeutic adjustment to target American Diabetes Association (ADA) criteria)
  Interventions: Drug: Cyclosporin; Behavioral: 'Diabetes Education / Management'
- Tacrolimus (Active Comparator): Patients receive tacrolimus (dose-adjusted to pre-established targets) as CNI and Diabetes Education / Management (therapeutic adjustment to target ADA criteria)
  Interventions: Drug: Tacrolimus; Behavioral: 'Diabetes Education / Management'

INTERVENTIONS:
Drug: Cyclosporin — Dose adjustment to pre-established targets
  Other Names: Neoral
  Arms: Cyclosporin
Drug: Tacrolimus — Dose adjustment to pre-established targets
  Other Names: Prograf
  Arms: Tacrolimus
Behavioral: 'Diabetes Education / Management' — therapeutic adjustment to target ADA criteria

SUMMARY:
Protocol Title: Randomized open label study comparing the metabolic control of first Kidney Transplant recipients with Type 2 Diabetes Mellitus (DM) receiving either Prograf or Neoral as part of a ATG induction, prednisone free and blood monitored Cellcept immunosuppressive regimen.

PURPOSE This is a single center medical research study to analyze post-transplant kidney recipients with pre-existing type 2 diabetes managed according to the recommended American Diabetes Association (ADA) guidelines. Prograf (Tac) and Neoral (CSA) are the two main medications to prevent rejection after transplantation. However, they may contribute to poorer diabetes control. The purpose of the study is to compare the effects of Prograf and Neoral on the control of Diabetes after kidney transplantation. In addition, all participants in this study will receive Thymoglobulin (anti-lymphocyte globulin) at the time of transplantation instead of long term prednisone (steroids).

DETAILED DESCRIPTION:
It has been accepted that patients with DM are associated with a greater risk of morbidity and mortality and hyperlipidemia, compromised graft function, stroke, nephropathy, atherosclerotic cardiovascular disease, graft-loss, infection, retinopathy, neuropathy, gastropathy, and vascular complications.2

Patients with pre-existing DM had a 1.9 times less survival days.3 In renal transplantation, twice as many patients with pre-existing diabetes die with functioning graft.4

DM has been shown to be predominantly the single most important predictor for adverse outcomes in terms of mortality and morbidity resulting from various end organ damages.

Poor DM control leads to an increased risk of both graft loss and patient death due to manifestations of end-stage DM.8 Chronic Allograft Nephritis (CAN) is a common finding at the 6th month post kidney transplant, especially in patients with blood glucose metabolism abnormalities.

Several conditions may lead the worsening of the diabetes after transplantation. First, for patients with ESRD the improvement of kidney function after kidney transplantation leads also to an increased clearance of circulating insulin. Second, most patients experience a significant improvement of well being after successful transplantation. Often their appetite is significantly improved, resulting in a significant weight gain - increasing insulin demand and resistance. Finally, most immunosuppressive medications are diabetogenic. Corticoid-steroids are well known for their strong diabetogenic effect and have been associated with post transplant diabetes. Calcineurin inhibitors are now the corner stone of immunosuppression for organ transplantation. This class of medication includes cyclosporine and tacrolimus. Both have been associated with post transplantation diabetes. Induction agents, including polyclonal antibodies (ex. Thymoglobulin) and monoclonal antibodies (ex. Anti Il-2 receptor, Zenapax, Simulect) are not found to cause hyperglycaemia. The two areas of possible intervention to minimize worse diabetes after transplantation are thus limited to 1) comprehensive diabetes education and 2) newer immunosuppressive regimen after transplantation.

1.1 Comprehensive Diabetes Education:

DM can arise both in the stressful time of organ failure or in the post-transplant phase. During a prospective study we conducted on solid organ transplant recipients with pre-existing and post transplant diabetes we observed the following trends:

* The complex nature of organ transplantation carries potential side effects, which are amenable to early intervention in the post transplant setting with patients who have diabetes through education and monitoring by the transplant team.
* Patients with poorly controlled diabetes post transplant have a higher incidence of post transplant morbidity.

Our study showed a 7% DM-related re-admissions within one year post-transplant for patients in the Diabetes and Transplant Program, compared to a 93% DM-related re-admission rate within one year for patients not enrolled in the Program.10

Further analysis of Stanford Medical Center's Transplant Diabetes Program revealed that patients' average HbA1c was 8.8% at intake into the program. Patients who were followed by this multi disciplinary Transplant Diabetes education team resulted in an average value of 7.2% following a minimum of three months of management. 11

1.2 Immunosuppression for Transplant Patients with Diabetes: The utilization of a calcineurin inhibitor in combination with steroids has contributed to the improved success of transplantation seen since the introduction of cyclosporine in 1983. Prograf, also a calcineurin inhibitor was introduce later (1989) and was associated with further improvement in results. Newer immunosuppressive medication has been introduced since then. There has been interest in the transplant community to use the new agents to achieve steroid minimization or avoidance. These strategies are very appealing for the diabetic patients as both steroids and calcineurin inhibitors are the most diabetogenic medication they receive after transplantation.

1.2.1 STEROIDS Stanford's Pediatric kidney transplant team have demonstrated the feasibility of steroid avoidance or rapid taper after kidney transplantation. Doctor Salvatierra team substituted Zenapax induction therapy for steroids in a series of pediatric kidney transplant recipients. Patients received as well tacrolimus and MMF for prophylaxis of rejection. They initially reported their experience with the first 34 patients (5-21 years old) treated with that protocol. The graft survival was 100 % and the incidence of acute rejection was rejection 6% compared with 15 % for historical controls receiving steroids. They had no post transplantation diabetes or high blood pressure, cholesterol was lower, obesity and appearance was also significantly better.12 Steroid avoidance is now the standard treatment for Stanford's Pediatric Transplant Program.

The adult Kidney Transplant Program has been able to reproduce the pediatric experience with a similarly designed steroid avoidance protocol. A slightly different approach has also been successfully used. Kidney transplant recipients received Thymoglobulin induction in lieu of Zenapax and received 4 small doses of steroids peri-operatively. So far 25 patients were treated with this minimal exposure to steroids. The graft and patient survival is 100% and only one episode of rejection was seen. This approach is preferred to the total avoidance of steroids since it is associated with a better initial kidney function.13 This later approach is currently used by Stanford's Adult Kidney Transplant Program for un-sensitized adult patients receiving a kidney transplant if they have a medical condition that could be exacerbated by the use of steroids; diabetes, obesity, osteopenia, and coronary artery disease.

Utilisation of Thymoglobulin was associated with a lower incidence of acute rejection than IL-2RA. Xiao et Al showed the absence of Post Transplant Diabetes Mellitus (PTDM) and decreased use of anti-hypertensive medication in the steroid free group.

Minimization of steroid use has clear metabolic benefits for the diabetic patients. Within Stanford University Transplant service there is enough experience to support its safe use. In this study, all patients will have minimal exposure to steroids. We have opted to give only peri-operative steroids (4 doses total) as in our experience this approach is associated with better initial graft function than the complete steroid avoidance. We also elected to use induction therapy with Thymoglobulin as it is associated with the lowest rate of rejection rate in the above mentioned studies.14

1.2.2 Calcineurin inhibitors Calcineurin inhibitors have also been associated with post transplant diabetes. The incidence of PTDM has been reported to be more than 30% depending on the calcineurin inhibitor used, (Cyclosporine vs. Prograf), trough level, race, and risk factors for diabetes all contribute to this number. These figures may underestimate the true incidence of PTDM, as most studies have not utilized the strict criteria of the ADA for diagnosis of diabetes. Most studies report a higher incidence of PTDM with the use of Prograf compared to Cyclosporine. The greater diabetogenicity of Prograf has been confirmed in a recent study investigating the new onset of diabetes both before and after kidney transplant.14 this study revealed that the incidence of new-onset diabetes was 70% higher in Prograf treated patients than with patients receiving Neoral.16 This contrasts with studies mentioned above where Prograf is used in steroid free protocols with no or very low incidence of post transplant diabetes.

Calcineurin inhibitors do remain the corner stone of immunosuppression at the present time, and even more so in the context of steroid minimization. It would thus be very important to determine if one of the two calcineurin inhibitors available on the market has a more favourable metabolic profile specifically for patients with pre-existing diabetes. Direct comparison between Neoral (micro-emulsion formulation of CSA) and Prograf has never been made in context of short steroid taper and specifically for non-insulin dependent diabetic patients.

Equitable comparison between Neoral and Prograf is difficult, as both drugs do not have the same pharmacokinetic profile. Trough (or pre-dose) level has been used to evaluate drug exposure and make dosage adjustment. Prograf has a more predictive correlation between the trough level and the total area under the curve (total drug exposure of the patient) than Neoral. C2 monitoring of CSA consists of measuring the drug level 2 hours after ingestion. The correlation of C2 monitoring of Neoral to the area under the curve is similar to the correlation of the trough for Prograf to the area under the curve (both R 2=0.92). C2 monitoring for Neoral has been associated with an increase in efficacy and reduction in toxicity. In this study we will use C2 monitoring for Neoral and trough monitoring for Prograf. Moderate minimization of the calcineurin inhibitor dosage will be used in this study in order to reduce the deleterious effect of the calcineurin inhibitors to the metabolism of glucose. A reduction of approximately 20% of our usual target level will be used.

1.2.3 Cellcept (MMF) Utilization of MMF is combination of Prograf or Neoral is the standard treatment after kidney transplantation. Mycophenolic acid (MPA) is the active component of MMF. Therapeutic drug monitoring of MPA has been shown to reduce rejection and toxicity.15 Furthermore; cyclosporine interferes with MPA metabolism resulting in a lower exposure to the drug compared to patients receiving Prograf when a fix dose is used. MPA monitoring may thus ensure that patients in our study are within therapeutic window of this immunosuppressive agent. This may prove to be even more crucial as they are not receiving steroids. MPA monitoring will also ensure that Neoral and Prograf groups receive the similar drug exposure to MPA.

1.2.4 Conclusion

Patients with diabetes are at higher risks of morbidity and mortality after kidney transplantation. Currently, there is no published data on the morbidity and mortality of these high risk patients from a prospective study that utilizes the American Diabetes Association (ADA) criteria for diabetes management and control, nor which addresses:

* The impact of steroids elimination on outcomes after kidney transplantation and metabolic control in patients with pre-existing type 2 diabetes.
* Optimization of CI therapy for post transplant patients with pre-existing type 2 DM and its impact on metabolic control.

The proposed study compares the effect of Calcineurin inhibitors have on metabolic control in the absence of corticosteroids to better optimize post-transplant patient outcomes and decrease morbidity in patients with DM. With close monitoring of transplant recipient immunosuppression protocol, elimination of CS and the reduction of CI therapy, we propose there will be a decrease in patient morbidity associated with DM.

The findings of this study may help:

* Identify optimal immunosuppression therapy for transplant patients with diabetes
* Decrease DM related co-morbidities and hospital readmissions
* Increase longevity of life and graft survival in transplant recipients with DM.
* Lower overall post-transplant health care costs that are attributed to the morbidity of immunosuppression therapy and diabetes.
* Promote better DM self-care in the transplant process
* Results from this study where 100% of the studied population is diabetic may provide further insight in the metabolism of glucose after transplantation resulting in better understanding of post transplant diabetes.

During the conduct of the study the outcomes were amended to included freedom from insulin therapy, estimated glomerular filtration rate (eGFR) as an indicator of graft function, post-operative survival up to 1 year, and biopsy-proven transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Patient is a recipient of a first cadaveric kidney, or a kidney living donor mismatched (at least one mismatch.)
2. Patient is a minimum of 18 years of age at the time of transplant.
3. Patient has type 2 non-insulin dependent diabetes.
4. Patient or legal guardian has signed and dated an Ethics Committee-approved informed consent document and is willing and able to follow study procedures.
5. If female and is childbearing potential, patient has a negative pregnancy test and utilizes adequate contraceptive methods.

Exclusion Criteria

1. Recipients of a transplant graft from a donor age 65 and older.
2. Recipient of a multi-organ transplant.
3. Patients who are being re-transplanted will not be eligible for study.
4. Patients who have lost a previous graft to rejection less than one year from transplant.
5. Patient has any form of substance abuse, psychiatric disorder, or a condition in the opinion of the investigator, may invalidate communication with the investigator.
6. PRA > 30%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Busque, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford university Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weir MR, Fink JC. Risk for posttransplant Diabetes mellitus with current immunosuppressive medications. Am J Kidney Dis. 1999 Jul;34(1):1-13. doi: 10.1016/s0272-6386(99)70101-0. PMID 10401009
- [Background] Sarwal MM, Yorgin PD, Alexander S, Millan MT, Belson A, Belanger N, Granucci L, Major C, Costaglio C, Sanchez J, Orlandi P, Salvatierra O Jr. Promising early outcomes with a novel, complete steroid avoidance immunosuppression protocol in pediatric renal transplantation. Transplantation. 2001 Jul 15;72(1):13-21. doi: 10.1097/00007890-200107150-00006. PMID 11468528
- [Background] Rigatto C. Clinical epidemiology of cardiac disease in renal transplant recipients. Semin Dial. 2003 Mar-Apr;16(2):106-10. doi: 10.1046/j.1525-139x.2003.16026.x. PMID 12641873
- [Background] Hamar P, Muller V, Kohnle M, Witzke O, Albrecht KH, Philipp T, Heemann U. Metabolic factors have a major impact on kidney allograft survival. Transplantation. 1997 Oct 27;64(8):1135-9. doi: 10.1097/00007890-199710270-00009. PMID 9355829
- [Background] Maes BD, Kuypers D, Messiaen T, Evenepoel P, Mathieu C, Coosemans W, Pirenne J, Vanrenterghem YF. Posttransplantation diabetes mellitus in FK-506-treated renal transplant recipients: analysis of incidence and risk factors. Transplantation. 2001 Nov 27;72(10):1655-61. doi: 10.1097/00007890-200111270-00014. PMID 11726827
- [Background] Revanur VK, Jardine AG, Kingsmore DB, Jaques BC, Hamilton DH, Jindal RM. Influence of diabetes mellitus on patient and graft survival in recipients of kidney transplantation. Clin Transplant. 2001 Apr;15(2):89-94. doi: 10.1034/j.1399-0012.2001.150202.x. PMID 11264633
- [Background] Gerber JC, Stewart DL. Prevention and control of hypertension and diabetes in an underserved population through community outreach and disease management: a plan of action. J Assoc Acad Minor Phys. 1998;9(3):48-52. PMID 9747058
- [Background] Navasa M, Bustamante J, Marroni C, Gonzalez E, Andreu H, Esmatjes E, Garcia-Valdecasas JC, Grande L, Cirera I, Rimola A, Rodes J. Diabetes mellitus after liver transplantation: prevalence and predictive factors. J Hepatol. 1996 Jul;25(1):64-71. doi: 10.1016/s0168-8278(96)80329-1. PMID 8836903

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclosporin: Patients receive cyclosporin (Neoral; dose-adjusted to pre-established targets) as immunosuppressive calcineurin inhibitor (CNI) and Diabetes Education / Management (therapeutic adjustment to target American Diabetes Association (ADA) criteria)
- Tacrolimus: Patients receive tacrolimus (Prograf; dose-adjusted to pre-established targets) as CNI and Diabetes Education / Management (therapeutic adjustment to target ADA criteria)
Period: Overall Study
Arm/Group | Cyclosporin | Tacrolimus
Started | 11 | 18
Completed | 9 | 5
Not Completed | 2 | 13

BASELINE CHARACTERISTICS:
Groups:
- Cyclosporin: Patients receive cyclosporin (dose-adjusted to pre-established targets) as CNI and Diabetes Education / Management (therapeutic adjustment to target ADA criteria)
- Total: Total of all reporting groups
Arm/Group | Cyclosporin | Tacrolimus | Total
Number analyzed (Participants) | 11 | 18 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 16 | 24
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 8 | 16 | 24

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Insulin Therapy Post Transplant
Description: The count of participants with freedom from insulin therapy post transplant is reported.
Time Frame: From hospital discharge to 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporin | Tacrolimus
Number analyzed (Participants) | 11 | 18
Participants | 3 | 4

2. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR) 1 Year Following Transplantation
Description: Values of ≥60 ml/min/1.73 m^2 are considered optimal; ≥30-59 ml/min/1.73 m^2 are indicative of successful graft function; lower values are indicative or graft dysfunction.
Time Frame: 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporin | Tacrolimus
Number analyzed (Participants) | 11 | 18
Participants
  ≥60 ml/min/1.73 m^2 | 4 | 6
  ≥30-59 ml/min/1.73 m^2 | 6 | 9
  <30 ml/min/1.73 m^2 | 1 | 3

3. Secondary Outcome: Patient Survival at One Year Post Transplantation
Description: Count of participants alive at one year post transplantation
Time Frame: Up to 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporin | Tacrolimus
Number analyzed (Participants) | 11 | 18
Participants | 10 | 16

4. Secondary Outcome: Count of Participants With Biopsy Proven Acute Rejection at One Year Post Transplantation
Time Frame: 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporin | Tacrolimus
Number analyzed (Participants) | 11 | 18
Participants | 1 | 3

ADVERSE EVENTS:
Arm/Group | Cyclosporin | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/18
Other Adverse Events (participants affected / at risk) | 0/11 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes